CLINICAL TRIAL: NCT03146663
Title: A Phase II Open-Label Study of NUC-1031 in Patients With Platinum-Resistant Ovarian Cancer
Brief Title: NUC-1031 in Patients With Platinum-Resistant Ovarian Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Despite promising efficacy and a good tolerability profile in Part I, it was decided not to initiate Part II as the pre-specified boundary for efficacy was uncertain to be met in this heavily pre-treated population with significant co-morbidities
Sponsor: NuCana plc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO-105; 2016-003287-39 (EudraCT Number)
Record Dates: First submitted 2017-05-04; First posted 2017-05-10 (Actual); Results first posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Ovarian Cancer
Keywords: Platinum-resistant; ovarian neoplasm; antineoplastic agents; ovarian diseases; cancer of the ovary
MeSH Terms: conditions — Ovarian Neoplasms; Ovarian Diseases | interventions — NUC-1031

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): NUC-1031 500 mg/m2 administered on Days 1, 8, and 15 of 28-day cycles
  Interventions: Drug: NUC-1031 500 mg
- Arm B (Experimental): NUC-1031 750 mg/m2 administered on Days 1, 8, and 15 of 28-day cycles
  Interventions: Drug: NUC-1031 750mg

INTERVENTIONS:
Drug: NUC-1031 500 mg — NUC-1031 500 mg/m2 on Days 1, 8, and 15 of a 28-day cycle.
  Other Names: fosgemcitabine palabenamide
  Arms: Arm A
Drug: NUC-1031 750mg — NUC-1031 750 mg/m2 on Days 1, 8, and 15 of a 28-day cycle
  Other Names: fosgemcitabine palabenamide
  Arms: Arm B

SUMMARY:
This study was designed to evaluate the effect of two dose levels of NUC-1031 (500 mg/m2 and 750mg/m2) in patients with ovarian cancer. The primary objective was to determine the anti-tumor activity of NUC-1031 at the selected dose level (500 mg/m2 or 750 mg/m2).

DETAILED DESCRIPTION:
A total of 53 patients were randomized, of whom 51 patients were treated in Part I of the study, 24 patients in the 500 mg/m2 arm and 27 patients in the 750 mg/m2 arm. Eligible, consenting patients received NUC-1031 by IV infusion on Days 1, 8, and 15 of each 28-day cycle. Patients continued to receive NUC-1031 until the occurrence of disease progression and underwent imaging every 8 weeks. After disease progression, patients were followed for overall survival.

Part II of the study was designed to select one of the treatment dose levels for further evaluation based on clinical and laboratory assessments of patients recruited in Part I. Despite promising efficacy and a good tolerability profile in Part I, it was decided not to initiate Part II as the pre-specified boundary for efficacy was uncertain to be met in this heavily pre-treated population with significant co-morbidities.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed written informed consent.
2. Original diagnosis and/or histological confirmation of high-grade serous, high-grade endometrioid, undifferentiated/unclassifiable epithelial ovarian, fallopian tube or primary peritoneal cancer.
3. Time from the last line of platinum-based chemotherapy of less than 6 months.
4. Received at least 3 prior chemotherapy-containing regimens.
5. Age ≥18 years.
6. Ability to comply with protocol requirements.
7. Patients are not of childbearing potential or they must agree to use a physical method of contraception.

Exclusion Criteria:

1. Disease that progressed while receiving initial line of platinum-based chemotherapy.
2. Received fewer than 3 prior chemotherapy-containing regimens.
3. Prior therapy with single-agent gemcitabine.
4. Prior history of hypersensitivity to gemcitabine.
5. Prior chemotherapy, radiation (other than short cycle of radiation to reduce bone pain), treatment with a VEGF inhibitor, PARP inhibitor or immunotherapy within 21 days of first receipt of study drug. Hormone therapy within 14 days of first receipt of study drug.
6. Residual side effects from chemotherapy or radiation, which have not gotten better except for nerve pain or tingling or hair loss.
7. Patients who have a history of another type of cancer diagnosed within the past 5 years, with the exception of adequately treated non-melanoma skin cancer curatively treated cervical cancer or ductal carcinoma in situ (DCIS) of the breast.
8. Presence of an serious illness, uncontrolled illness, or active infection requiring IV antibiotics.
9. Presence of any serious illnesses, serious medical conditions, serious medical history, active bacterial or viral infections including hepatitis B or C, or known to be HIV positive.
10. Currently pregnant, lactating or breastfeeding.
11. History of blocked intestines because of ovarian cancer, unless fully resolved.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2017-09-28 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Oelmann, MD PhD, Study Director — NuCana plc
Locations (17):
- United States (10):
  - Arizona Oncology Associates, PC - HAL, Phoenix, Arizona
  - Arizona Oncology Associates, PC - HOPE, Tucson, Arizona
  - Rocky Mountain Cancer Centers, LLP, Lakewood, Colorado
  - Florida Cancer Specialists and Research Institute, St. Petersburg, Florida
  - Minnesota Oncology Hematology, P.A., Edina, Minnesota
  - SCRI - HCA Health Midwest, Kansas City, Missouri
  - Nashville Tennessee Oncology, Nashville, Tennessee
  - Texas Oncology - South Austin, Austin, Texas
  - Texas Oncology The Woodlands, Gynecologic Oncology, The Woodlands, Texas
  - Texas Oncology - Tyler, Tyler, Texas
- United Kingdom (7):
  - Edinburgh Cancer Centre, Edinburgh
  - Cancer Research UK Clinical Trial Unit, Glasgow
  - St Bartholomew's Hospital, London
  - University College London Hospital, London
  - Royal Marsden Hospital, London
  - Imperial College Healthcare NHS Trust, London
  - Oxford University Hospital Foundation Trust, Oxford

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 87 patients were screened, of whom 53 patients were randomized and 51 patients received at least one dose of NUC-1031. These 51 patients were included in the full analysis set and the safety analysis set.
Pre-assignment Details: Screening details: Patients with histologically-confirmed platinum-resistant high-grade serious, high-grade endometrioid, epithelial cancer of the ovary, fallopian tube or primary peritoneum (here termed 'ovarian cancer'), who had been treated with 3 or more prior chemotherapy regimens were eligible. The Screening visit was to occur within 28 days of Cycle 1 Day 1.
Period: Overall Study
Arm/Group | Arm A | Arm B
Started | 25 | 28
Completed | 24 | 27
Not Completed | 1 | 1
Not completed — Did not receive study treatment | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 25 | 28 | 53
Age, Customized [Count of Participants; unit: Participants]
  <55 years | 6 | 4 | 10
  55 - <66 years | 6 | 10 | 16
  66 - 75 years | 9 | 10 | 19
  >75 years | 4 | 4 | 8
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 25 | 28 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 24 | 28 | 52
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 0 | 1
  Black/African American | 0 | 2 | 2
  White | 23 | 26 | 49
  Other | 1 | 0 | 1
Original diagnosis [Count of Participants; unit: Participants]
  Ovarian | 16 | 20 | 36
  Fallopian tube | 4 | 2 | 6
  Primary peritoneal | 3 | 5 | 8
  Other | 2 | 0 | 2
  Not recorded | 0 | 1 | 1
Metastatic disease [Count of Participants; unit: Participants]
  Yes | 25 | 26 | 51
  No | 0 | 1 | 1
  Not recorded | 0 | 1 | 1
Time since initial diagnosis [Median (Full Range); unit: years] — Population: Time since initial diagnosis for one patient in Arm B (750 mg/m2) was unknown.
  years
    number analyzed (Participants) | 25 | 27 | 52
    (all) | 4.3 [1.8 to 17.3] | 5.6 [1.7 to 15.6] | 5.0 [1.7 to 17.3]
Histology [Count of Participants; unit: Participants]
  High grade serous | 24 | 23 | 47
  High grade endometroid | 1 | 1 | 2
  Other | 0 | 3 | 3
  Not recorded | 0 | 1 | 1
Stage at screening [Count of Participants; unit: Participants] — Ovarian cancer stages range from Stage I-IV, classifying how much cancer is in the body. The lower the number, the less the cancer has spread through the body and the higher the number the more the cancer has spread. Stage I-III cancer is present with the higher the number the larger the tumour and the more it has spread into nearby tissues; Stage IV cancer has spread to distant parts of the body. Stage is determined using the FIGO (International Federation of Gynecology and Obstetrics) system or the AJCC (American Joint Committee on Cancer) TNM staging system.
  Participants
    Stage I | 1 | 0 | 1
    Stage II | 1 | 0 | 1
    Stage III | 8 | 7 | 15
    Stage IV | 13 | 18 | 31
    Unknown | 2 | 2 | 4
    Not recorded | 0 | 1 | 1
Documented deleterious BRCA mutation [Count of Participants; unit: Participants]
  Yes | 4 | 4 | 8
  No | 21 | 23 | 44
  Unknown | 0 | 1 | 1
Eastern Cooperative Oncology Group (ECOG) performance status [Count of Participants; unit: Participants] — ECOG is a scale (0-5) and criteria used to assess a patient's performance or functional status. 0 = fully active (best), able to carry on all pre-disease performance without restriction; 1=restricted in physically strenuous activity, but ambulatory and able to carry out light or sedentary work; 2 = ambulatory (≥50% waking hours), capable of all selfcare but unable to carry out work activities; 3 = capable of only limited selfcare and confined to bed or chair ≥50% waking hours; 4 = completely disabled, cannot carry on selfcare, totally confined to bed or chair; 5 = dead (worst).
  Participants
    0 | 8 | 12 | 20
    1 | 16 | 16 | 32
    Unknown | 1 | 0 | 1
Comorbidity at baseline [Count of Participants; unit: Participants]
  Yes | 19 | 19 | 38
  No | 6 | 9 | 15
Prior systemic cancer therapy [Count of Participants; unit: Participants]
  Yes | 24 | 27 | 51
  No | 1 | 1 | 2
Time to progression after start of most recent chemotherapy [Count of Participants; unit: Participants]
  <= 1 month | 0 | 0 | 0
  >1 to 6 months | 14 | 15 | 29
  >6 to 9 months | 2 | 1 | 3
  >9 to 12 months | 1 | 0 | 1
  >12 months | 1 | 0 | 1
  Missing | 7 | 12 | 19
Treatment-free interval from completion of most recent chemotherapy [Count of Participants; unit: Participants]
  <= 1 month | 2 | 3 | 5
  >1 to 3 months | 14 | 10 | 24
  >3 to 6 months | 5 | 9 | 14
  >6 to 9 months | 2 | 4 | 6
  >9 months | 1 | 1 | 2
  Missing | 1 | 1 | 2
Number of prior lines of therapy [Median (Full Range); unit: Therapies] | 4.5 [3 to 12] | 5.0 [3 to 11] | 4.8 [3 to 12]
Prior gemcitabine-containing regimen [Count of Participants; unit: Participants]
  Yes | 13 | 17 | 30
  No | 12 | 11 | 23

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response
Description: Best overall response to study treatment, as assessed by blinded independent central review according to RECIST v1.1, in the evaluable population of patients who received at least one dose of study treatment and had measurable disease at baseline.
  Complete Response (CR): disappearance of all target and non-target lesions, normalization of tumor markers, and pathological lymph nodes must have short axis measurements <10 mm.
  Partial Response (PR): ≥30% decrease in the sum of measures of target lesions, taking as reference the baseline sum of diameters. Non-target lesions must be non-progressive disease.
  Stable Disease (SD): neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as reference the smallest sum of diameters on study.
  Progressive Disease (PD): ≥20% increase in the sum of measured lesions taking as reference the smallest sum of diameters recorded on study and an absolute increase of ≥5mm.
Time Frame: Assessed from date of randomization until disease progression, up to end of the study (approximately 2 years)
Population: Evaluable population are patients who received at least one dose of study treatment and who had measurable disease at baseline.
Measure: Count of Participants; unit: Participants
Groups:
- Arm B: NUC-1031 750 mg/m2 administered on Days 1, 8 and 15, of 28-day cycles
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 24 | 26
Participants
  Complete response | 0 | 1
  Partial response | 2 | 0
  Stable disease | 8 | 8
  Progressive disease | 12 | 10
  Not evaluable | 1 | 2
  Missing | 1 | 5

2. Post Hoc Outcome: Best Overall Response (in Evaluable for Response Set)
Description: Post-hoc analysis of best overall response to study treatment, as assessed by blinded independent central review according to RECIST v1.1, in the per protocol evaluable for response set of patients. Per protocol evaluable for response set is defined as all patients from the Full Analysis Set who had measurable disease at baseline, at least one post-baseline scan and who received a dose of NUC-1031 on all dosing days of Cycle 1.
Time Frame: Assessed from date of randomization until disease progression, up to end of the study (approximately 2 years)
Population: Reporting group
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 17 | 5
Participants
  Complete response | 0 | 1
  Partial response | 2 | 0
  Stable disease | 6 | 1
  Progressive disease | 8 | 3
  Not evaluable | 1 | 0

ADVERSE EVENTS:
Time Frame: Date of consent until 30 days after the last dose of study treatment, up to end of the study (approximately 2 years)
Arm/Group | Arm A | Arm B
All-Cause Mortality (participants affected / at risk) | 21/24 | 21/27
Serious Adverse Events (participants affected / at risk) | 8/24 | 10/27
Other Adverse Events (participants affected / at risk) | 24/24 | 26/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=24) | Arm B (N=27)
Vomiting (Gastrointestinal disorders) | 2 | 2
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Infection (Infections and infestations) | 1 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection bacterial (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Pyrexia (General disorders) | 1 | 1
Asthenia (General disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Super vena cava syndrome (Vascular disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=24) | Arm B (N=27)
Nausea (Gastrointestinal disorders) | 16 (18) | 15 (24)
Vomiting (Gastrointestinal disorders) | 12 (13) | 12 (13)
Diarrhoea (Gastrointestinal disorders) | 10 (14) | 5 (7)
Constipation (Gastrointestinal disorders) | 8 (9) | 5 (8)
Abdominal Pain (Gastrointestinal disorders) | 5 (7) | 5 (7)
Abdominal distension (Gastrointestinal disorders) | 4 (4) | 1 (2)
Ascites (Gastrointestinal disorders) | 3 (3) | 1 (1)
Fatigue (General disorders) | 16 (27) | 14 (23)
Pyrexia (General disorders) | 7 (9) | 2 (4)
Oedema peripheral (General disorders) | 2 (4) | 4 (5)
Alanine aminotransferase increased (Investigations) | 7 (10) | 6 (7)
Aspartate aminotransferase increased (Investigations) | 6 (8) | 5 (7)
Neutrophil count decreased (Investigations) | 2 (2) | 6 (14)
Blood alkaline phosphatase increased (Investigations) | 3 (4) | 2 (2)
White blood cell count decreased (Investigations) | 3 (4) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 8 (12) | 6 (9)
Thrombocytopaenia (Blood and lymphatic system disorders) | 5 (6) | 5 (9)
Neutropaenia (Blood and lymphatic system disorders) | 6 (12) | 3 (8)
Decreased appetite (Metabolism and nutrition disorders) | 7 (9) | 6 (9)
Dehydration (Metabolism and nutrition disorders) | 5 (6) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 4 (4)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2)
Dizziness (Nervous system disorders) | 3 (3) | 4 (6)
Headache (Nervous system disorders) | 4 (7) | 2 (2)
Urinary tract infection (Infections and infestations) | 4 (9) | 2 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Vision blurred (Eye disorders) | 3 (3) | 1 (2)
Dysuria (Renal and urinary disorders) | 3 (4) | 0 (0)
Tachycardia (Cardiac disorders) | 3 (3) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 2 (3)
Abdominal pain lower (Gastrointestinal disorders) | 2 (2) | 1 (1)
Asthenia (General disorders) | 2 (2) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 2 (2)
Influenza like illness (General disorders) | 2 (2) | 1 (1)
Mucosal inflammation (General disorders) | 2 (2) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 2 (2) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Dysgeusia (Nervous system disorders) | 2 (2) | 2 (2)
Lethargy (Nervous system disorders) | 2 (2) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1)

LIMITATIONS AND CAVEATS:
Despite promising efficacy and a good tolerability profile in Part I, it was decided not to initiate Part II as the pre-specified boundary for efficacy was uncertain to be met in this heavily pre-treated population with significant co-morbidities.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-10-11): https://cdn.clinicaltrials.gov/large-docs/63/NCT03146663/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-26): https://cdn.clinicaltrials.gov/large-docs/63/NCT03146663/SAP_001.pdf